CLINICAL TRIAL: NCT04885764
Title: Profiling Antibody Status and Vaccine Effectiveness in Post Vaccination With SARS CoV2 in Ain Shams University
Acronym: ASU-VAC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Samia Girgis, Professor of Clinical Pathology, Faculty of Medicine, Ain Shams University, Cairo, Egypt, Ain Shams University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU P01b / 2021
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Covid19
Keywords: Egypt; Ain Shams University; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Astrazeneca/Oxford Vaccine — Viral non replicated vector vaccine contains the gene that encodes for the spike protein on the surface of the SARS-CoV-2 virus given Intramuscular injection in 2 doses 3 months apart
  Other Names: Vaxzevria
Biological: Sinopharm vaccine — Inactivated vaccine given intramuscular injection in 2 doses 3 weeks apart

SUMMARY:
This is a prospective intervention study to assess the effectiveness of both the live attenuated and messenger RNA vaccines against SARS-CoV-2 infection

DETAILED DESCRIPTION:
This is a prospective intervention study to assess the short-term effectiveness of the first dose of both the live attenuated and messenger RNA vaccines against SARS-CoV-2 infection by monitoring the antibodies (IgG, IgM and level of neutralizing antibodies) in sera of post-vaccinated persons.

The study also will monitor the incidence of SARS-CoV-2 infection among vaccinees just before the first dose administration, 3 weeks after immunization, at the administration of the second dose, 14 days following the second dose and after 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Candidate for receiving vaccination according to health care authorties prioritaizaton

Exclusion Criteria:

1. SARS-CoV-2 recovered cases <3 months
2. Individuals who are currently infected with Sars-COV-2 and/or with respiratory symptoms with fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Short-term effectiveness | 21 days of the first dose of vaccine
  Assess the short-term effectiveness of the first dose of both the live attenuated and messenger RNA vaccines against SARS-CoV-2 infection by monitoring the antibodies (IgG, IgM and level of neutralizing antibodies) in sera of postvaccinated persons three weeks after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Samia E Girgis, M.D, Principal Investigator — Faculty of Medicine Ain Shams University
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: Undecided